CLINICAL TRIAL: NCT03605979
Title: Continuous Glucose Monitoring and Hypoglycemia Unawareness in Type 1 Diabetes: a Pilot Study
Brief Title: Continuous Glucose Monitoring and Hypoglycemia Unawareness in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2017Ao003
Record Dates: First submitted 2018-07-19; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; hypoglycemia unawareness; Insulin pump; Continuous glucose monitoring systems; Low glucose suspend
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetes group: Patient with hypoglycemia unawareness

SUMMARY:
Looking for strict normoglycemia in type 1 diabetes increases the risk of hypoglycemia, exposing to hypoglycemia unawareness. It has been shown that the early correction of hypoglycemia can help recovering the perception of hypoglycemia. The purpose of this prospective study was to assess the value of sensor-augmented insulin-pump therapy to treat hypoglycemia unawareness.

DETAILED DESCRIPTION:
To confirm hypoglycemia unawareness, patients answered a questionnaire based on the items explored by the model of Clarke 19 about hypoglycemia and hypoglycemia awareness. The eligibility of patients was confirmed by a blinded CG M recording using the trademark iPro ™ 2 sensor for 6 days. During this period the patient reported on a logbook the perception of their hypoglycemia, symptoms and how any hypoglycemia was corrected. Hypoglycemic manifestations were divided into adrenergic (shakiness, anxiety, palpitations, sweating, hunger, nausea, headache, coldness and pallor) and neuroglycopenic effects (impaired judgment, moodiness, paresthesia, emotional lability, confusion, ataxia, double vision, amnesia, seizures and lethargy). The confrontation of hypoglycemia detected by the blinded CG M and self-reported hypoglycemia validated the diagnosis of hypoglycemia unawareness.

Patients used the Paradigm® Veo™ pump and glucose sensors (trademark : Enlite®) with an hypoglycemia alarm set at sensor glucose value of 70 mg/dL while the LG S option was set to suspend insulin delivery at a sensor glucose value of 50 mg/dL or less. These thresholds allowed an active correction of hypoglycemia by the patient between 50 and 70 mg/dL. Patients were educated to use the system and to treat and manage hypoglycemia. Pump data were uploaded using the trademark Medtronic CareLink™ Management Software for Diabetes during visits at 10 days (D10), 2 months (M2) and 3 months (M3). Hypoglycemia awareness was assessed by an initial quiz that was repeated at M3 and 6 months (M6). A blinded CGM iPro ™ 2 was also realized at M3 to validate the modifications after sensor-augmented insulin-pump therapy.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* type 1 diabetes
* had been treated with insulin pump for more than three months
* had hypoglycemia unawareness with a hypoglycemia perception threshold below 60 mg/dL and/or had had at least one severe hypoglycemia event in the previous year

Exclusion Criteria:

* > 18 years
* any serious disease that could interfere with the study
* pregnancy,
* incompatibility with monitoring,
* irregular management of diabetes,
* hearing loss and low vision,
* preventing them from using the devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hypoglycemia unawareness
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2013-02-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Glycemia measured by continuous glucose monitoring (CGM) and pump | Day 0
Glycemia measured by continuous glucose monitoring (CGM) and pump | day 10
Glycemia measured by continuous glucose monitoring (CGM) and pump | Month 2
Glycemia measured by continuous glucose monitoring (CGM) and pump | Month 3

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Zalzali M, Houdelet-Guerinot V, Socquard E, Thierry A, Delemer B, Lukas-Croisier C. Continuous glucose monitoring and hypoglycemia unawareness in type 1 diabetes: a pilot study. Minerva Endocrinol. 2017 Sep;42(3):195-202. doi: 10.23736/S0391-1977.16.02326-9. Epub 2015 Jul 10. PMID 26159765